CLINICAL TRIAL: NCT01446965
Title: Vest Prevention of Early Sudden Death Trial: Prevention of Sudden Death After Myocardial Infarction Using a LifeVest Wearable Cardioverter-defibrillator (Formerly VEST/PREDICTS)
Brief Title: Vest Prevention of Early Sudden Death Trial and VEST Registry
Acronym: VEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90D0114; NCT00628966 (obsolete NCT alias)
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Results first posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-12

CONDITIONS: Myocardial Infarction; Ventricular Dysfunction; Sudden Death; Ventricular Tachycardia; Ventricular Fibrillation
Keywords: myocardial infarction, acute; myocardial infarction; ventricular dysfunction; death, sudden, cardiac; death, sudden; death; ventricular tachycardia; ventricular fibrillation; defibrillation, electric; cardioversion, electric; electric countershock; defibrillators, external
MeSH Terms: conditions — Myocardial Infarction; Ventricular Dysfunction; Death, Sudden; Tachycardia, Ventricular; Ventricular Fibrillation; Death, Sudden, Cardiac; Death

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wearable defibrillator (Experimental): subjects in the Device Group will receive a LifeVest® wearable cardioverter-defibrillator (manufacturer: ZOLL Medical Corporation) plus guideline-directed medical therapy for post-myocardial infarction patients
  Interventions: Device: wearable defibrillator
- Conventional treatment (No Intervention): subjects in the Control Group will only receive guideline-directed medical therapy for post-myocardial infarction patients

INTERVENTIONS:
Device: wearable defibrillator — LifeVest wearable defibrillator
  Other Names: LifeVest; wearable cardioverter-defibrillator; WCD; WD
  Arms: Wearable defibrillator

SUMMARY:
This study explores the hypothesis that wearable defibrillators can impact mortality by reducing sudden death during the first three months after a heart attack in persons with high risk for life-threatening arrhythmias.

DETAILED DESCRIPTION:
In patients with ventricular dysfunction immediately following myocardial infarction, sudden death may be responsible for up to 50% of total mortality. Wearable defibrillators may reduce sudden death by providing immediate detection and treatment of ventricular arrhythmias. This study is design to demonstrate a reduction in sudden death measured at three months following myocardial infarction among patients who have ventricular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients identified in the hospital or within 7 days after discharge with a diagnosis of an acute MI (STEMI or Non-STEMI)
* LV ejection fraction ≤35% determined at the following time point:

  1. If no PCI within the first 8 hours following the MI: ≥ 8 hours after MI
  2. If acute PCI occurs within 8 hours of MI: ≥8 hours after PCI
  3. If CABG is planned (before or within 7 days of discharge), wait to enroll and then use the most recent assessment at least 48 hours post CABG
* Age ≥ 18 years

Exclusion Criteria:

* Existing ICD or indication for an ICD at the time of screening
* Existing unipolar pacemakers/leads
* Chronic renal failure requiring hemodialysis after hospital discharge
* Chest circumference too small or too large for LifeVest garment*
* Participants discharged to an institutional setting with an anticipated stay > 7 days
* Pregnancy
* Inability to consent
* Any other condition or circumstance that in the judgment of the clinician makes the participant unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2348 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey E Olgin, MD, Principal Investigator — University of California, San Francisco; Byron K Lee, MD, Study Director — University of California, San Francisco; Mark J Pletcher, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (71):
- United States (57):
  - Alaska Heart Institute, Anchorage, Alaska
  - Cardiovascular Consultants Heart Center, Fresno, California
  - Salinas Valley Memorial Healthcare System, Salinas, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Christiana Care Health Services, Newark, Delaware
  - University of Florida, Gainesville, Florida
  - Watson Clinic for Research, Inc., Lakeland, Florida
  - Melbourne Cardiac Resarch Institute, Melbourne, Florida
  - Florida Heart Group/Florida Hospital, Orlando, Florida
  - Advocate Christ Hospital, Oak Lawn, Illinois
  - Lutheran General, Park Ridge, Illinois
  - The Heart Group/Deaconess Hospital, Evansville, Indiana
  - Indiana University, Indianapolis, Indiana
  - St. Vincent Medical Group, Indianapolis, Indiana
  - Western Kentucky Heart and Lung, Bowling Green, Kentucky
  - University of Kentucky Gill Heart Institute, Lexington, Kentucky
  - Ochsner Clinic, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial, Worcester, Massachusetts
  - The Valley Hospital, Ridgewood, New Jersey
  - Presbyterian Heart Group, Albuquerque, New Mexico
  - Albany Associates in Cardiology, Albany, New York
  - United Health Services, Johnson City, New York
  - Long Island Jewish Hospital, New Hyde Park, New York
  - St. Luke's- Roosevelt Hospital Center, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Huntington Hospital, New York, New York
  - University Cardiovascular Associates (Rochester), Rochester, New York
  - Stony Brook University, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina @ Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Heart Research, Raleigh, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University Hospital Case Medical Center, Columbus, Ohio
  - North Ohio Heart Center-North Ohio Research, Elyria, Ohio
  - Cardiovascular Research Center, LLC/Mercy St Vincent, Toledo, Ohio
  - Oklahoma Heart Institute-Hillcrest, Tulsa, Oklahoma
  - Oregon Heart & Vascular, Springfield, Oregon
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Geisinger Heart Institute, Danville, Pennsylvania
  - The Guthrie Clinic/Guthrie Medical Group, Sayre, Pennsylvania
  - Brown Medical School-Rhode Island Hospital, Providence, Rhode Island
  - Providence/South Carolina Heart Center, Columbia, South Carolina
  - McLeod Health/Pee Dee Cardiology, Florence, South Carolina
  - Wellmont Holston Valley, Kingsport, Tennessee
  - Turkey Creek Medical Center, Knoxville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Carilion Clinic, Roanoke, Virginia
  - Cardiac Study Center, Tacoma, Washington
- Germany (7):
  - Med. Uniklinik Heidelberg, Heidelberg, Deutschland
  - Herzzentrum Duisburg Kaiser-Wilhelm-Krankenhaus, Duisburg, North Rhine-Westphalia
  - Klinikum Links der Weser gGmbh Klinik, Bremen
  - Klinikum Göttingen Georg-August-Universität Göttingen, Göttingen
  - Klinikum der Stadt Ludwigshafen, Ludwigshafen
  - UNIVERSITÄTSMEDIZIN der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Mannheim, Mannheim
- Poland (7):
  - Gdanski Uniwersytet Medyczny, Gdansk
  - Specjalistyczna Poradnia Kardiologiczna, Kielce
  - Mc Tronik, Lodz
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Ministerstwa Spraw Wewnetrznych w Rzeszowie, Rzeszów
  - II Klinika Choroby Wiencowej, Instytut Kardiologii (Institute of Cardiology, Clinic II), Warsaw
  - Medical University of Warsaw, Warsaw
  - Institute of Cardiology, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Olgin JE, Pletcher MJ, Vittinghoff E, Wranicz J, Malik R, Morin DP, Zweibel S, Buxton AE, Elayi CS, Chung EH, Rashba E, Borggrefe M, Hue TF, Maguire C, Lin F, Simon JA, Hulley S, Lee BK; VEST Investigators. Wearable Cardioverter-Defibrillator after Myocardial Infarction. N Engl J Med. 2018 Sep 27;379(13):1205-1215. doi: 10.1056/NEJMoa1800781. PMID 30280654
- See also: Linked to VEST/PREDICTS registration: NCT00628966 — https://clinicaltrials.gov/show/NCT00628966

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2008 through April 2017, the investigators enrolled 2348 participants at 76 sites in the United States, at 24 in Poland, at 6 in Germany, and at 2 in Hungary. One U.S. site was dismissed on June 24, 2014, and the 46 participants at that site were excluded from the analyses, due to irregularities found by the institutional review board at the site. Thus, a total of 2302 participants were included in the analyses (1524 participants in the device group and 778 in the control group).
Groups:
- Wearable Defibrillator: subjects in the Device Group will receive a LifeVest® wearable cardioverter-defibrillator (WCD) (manufacturer: ZOLL Medical Corporation) plus guideline-directed medical therapy for post-myocardial infarction patients
  wearable defibrillator: LifeVest wearable defibrillator
Period: Randominization
Arm/Group | Wearable Defibrillator | Conventional Treatment
Started | 1554 | 794
Completed | 1524 | 778
Not Completed | 30 | 16
Not completed — One site was dismissed due to IRB irregularity | 30 | 16
Period: Participants Followed and Analyzed
Arm/Group | Wearable Defibrillator | Conventional Treatment
Started | 1524 | 778
Received WCD | 1481 | 0
Never Wore WCD (n=43 participants in the treatment group withdrew consent prior to receiving WCD or refused WCD fitting) | 43 | 0
Never Given WCD | 0 | 758
Given WCD Out of Protocol (n=20 participants in the control group received WCD by prescription outside of protocol by treating physician) | 0 | 20
Completed | 1514 | 766
Not Completed | 10 | 12
Not completed — Lost to Follow-up | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wearable Defibrillator | Conventional Treatment | Total
Number analyzed (Participants) | 1524 | 778 | 2302
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (12.6) | 61.4 (12.4) | 61.2 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex data not available for all randomized
  Participants
    number analyzed (Participants) | 1521 | 772 | 2293
    Female | 413 | 195 | 608
    Male | 1108 | 577 | 1685
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 25 | 12 | 37
  Asian | 23 | 14 | 37
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 143 | 75 | 218
  White | 1279 | 636 | 1915
  More than one race | 20 | 14 | 34
  Unknown or Not Reported | 33 | 27 | 60
Left ventricular ejection fraction [Mean (Standard Deviation); unit: percentage of total amount of blood] — Left ventricular ejection fraction is reported as percent of the total amount of blood in the left ventricle pushed out with each heartbeat. An ejection fraction of 35 percent or less was an inclusion criterion for the study.
  percentage of total amount of blood | 28.2 (6.1) | 28.2 (5.8) | 28.2 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Sudden Death Mortality
Description: For witnessed deaths, sudden cardiac death will be defined as an unexpected non-traumatic, non-self-inflicted fatality in otherwise stable participants who die within one hour of the onset of the terminal symptoms. For unwitnessed deaths, participants will meet the definition of sudden death if they are found dead within 24 hours of being well, assuming there is no evidence of another cause of death during that time period.
Time Frame: three months after myocardial infarction
Population: A total of 2302 participants were included in the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Wearable Defibrillator | Conventional Treatment
Number analyzed (Participants) | 1524 | 778
Participants | 25 | 19

2. Secondary Outcome: All Cause Mortality
Description: All deaths, due to any cause
Time Frame: three months after myocardial infarction
Measure: Count of Participants; unit: Participants
Arm/Group | Wearable Defibrillator | Conventional Treatment
Number analyzed (Participants) | 1524 | 778
Participants | 48 | 38

3. Secondary Outcome: Compliance With Wearable Defibrillator Use
Description: daily wear time of the device
Time Frame: three months after myocardial infarction
Population: Conventional treatment participants did not wear defibrillator.
Measure: Median (Inter-Quartile Range); unit: hours per day
Arm/Group | Wearable Defibrillator | Conventional Treatment
Number analyzed (Participants) | 1524 | 0
hours per day | 18 [3.8 to 22.7] |

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Wearable Defibrillator | Conventional Treatment
All-Cause Mortality (participants affected / at risk) | 48/1524 | 38/778
Serious Adverse Events (participants affected / at risk) | 475/1524 | 253/778
Other Adverse Events (participants affected / at risk) | 1421/1524 | 714/778
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wearable Defibrillator (N=1524) | Conventional Treatment (N=778)
CHD hospitalization, 1st event post-randomization (Cardiac disorders) | 475 (475) | 253 (253)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Wearable Defibrillator (N=1524) | Conventional Treatment (N=778)
Fatigue (General disorders) | 510 | 274
Back pain (Musculoskeletal and connective tissue disorders) | 283 | 137
Trouble sleeping (General disorders) | 551 | 264
Dizziness (General disorders) | 344 | 166
Fainting (General disorders) | 59 | 36
Nausea (Gastrointestinal disorders) | 132 | 85
Headache (General disorders) | 259 | 136
Palpitations (Cardiac disorders) | 327 | 182
Chest pain (Cardiac disorders) | 265 | 151
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 548 | 321
Rash in any location (Skin and subcutaneous tissue disorders) | 216 | 50
Rash on torso (Skin and subcutaneous tissue disorders) | 184 | 27
Itch in any location (Skin and subcutaneous tissue disorders) | 243 | 45
Itch on torso (Skin and subcutaneous tissue disorders) | 205 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT01446965/Prot_SAP_000.pdf